CLINICAL TRIAL: NCT04948957
Title: Changes in Cerebral Oxygenation and Cognitive Functions During Controlled Hypotension
Brief Title: Changes in Cerebral Oxygenation and Cognitive Functions
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Bengü Gülhan Aydin, Associate Professor, Zonguldak Bulent Ecevit University
Other Study IDs: 2013-81-03/09
Record Dates: First submitted 2021-06-12; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Hypotension; Controlled; Cognitive Dysfunction
Keywords: cerebral oxygenation; cognitive function; esmolol; nitroglycerine
MeSH Terms: conditions — Hypotension; Cognitive Dysfunction | interventions — esmolol; Nitroglycerin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- esmolol (Group E)
  Interventions: Drug: Esmolol
- nitroglycerin (Group N)
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Esmolol
  Groups: esmolol (Group E)
Drug: Nitroglycerin
  Groups: nitroglycerin (Group N)

SUMMARY:
The present study aimed to assess the influence of nitroglycerin and esmolol-induced hypotension on cerebral oxygen saturation by using near-infrared spectroscopy and postoperative cognitive function in patients undergoing nasal surgery.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* patients with ASA physical status of I-II
* aged 18-65 years

Exclusion Criteria:

* Age under 18 or above 65
* ASA > II
* coagulation disorders
* history of cardiovascular and cerebrovascular disease
* poor Blood Pressure control
* anemia, pregnancy, addiction to opioids
* body mass index (BMI) > 35
* intraoperative systolic BP < 65 mmHg
* surgical duration less than 30 minutes or more than 160 minutes
* need for an intraoperative sympathomimetic drug and the use of other hypotensive drugs
* preoperative Mini-Mental State Examination (MMSE) score of 23 or less.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - required controlled hypotension scheduled for nasal surgeries
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
effects of controlled hypotension on cerebral oxygen saturation | until end of the surgical procedure.
  influence of nitroglycerin and esmolol-induced hypotension on cerebral oxygen saturation by measuring regional cerebral oxygen saturation using Near-Infrared Spectroscopy

SECONDARY OUTCOMES:
effects of controlled hypotension on cognitive function | 24 hour before surgery and 24 hour after surgery
  influence of nitroglycerin and esmolol-induced hypotension on postoperative cognitive function using mini mental test score

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes